CLINICAL TRIAL: NCT05382611
Title: miRNA in Patients With Thoracic, Abdominal and Intracranial Aneurysms
Acronym: miRNA
Status: Completed | Type: Observational
Sponsor: Na Homolce Hospital (Other)
Collaborators: Czech Academy of Sciences (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Miroslav Prucha, M.D., PhD., Assoc.Prof, Na Homolce Hospital
Other Study IDs: IG144101
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Vascular Aneurysm
Keywords: miRNA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Aneurysmatic tissue, healthy tissue and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients Controls: Control group
  Interventions: Diagnostic Test: ngs next generation sequencing
- Patients with aneurysma: Patients with aneurysma
  Interventions: Diagnostic Test: ngs next generation sequencing

INTERVENTIONS:
Diagnostic Test: ngs next generation sequencing — the samples from aneurysmatic tissue and healthy aortic tissue will be investigated using NGS

SUMMARY:
To assess the expression of miRNA in patients with TAA, AAA in aneurysmatic tissue and to compare this expression with the healthy tissue in the same patient.

In the same cohort, to asses the presence of miRNA in plasma and to compare with the control group.

Over the period of three years,to follow subjects in order to assess if the presence of certain miRNAs speeds up or slows down the progression of disease.

In patients with intracranial aneurysms to detect miRNA in plasma especially in patients with familial occurrence.

DETAILED DESCRIPTION:
MicroRNAs constitute a recently discovered class of non-coding RNAs that play key roles in the regulation of gene expression. Acting at the post-transcriptional level, MicroRNAs have been shown to be involved in a wide range of biological processes such as cell cycle control, apoptosis and several developmental and physiological processes including stem cell differentiation, hematopoiesis, hypoxia, cardiac and skeletal muscle development. In addition to their important roles in healthy individuals, microRNAs have also been implicated in a number of diseases including a broad range of cancers, cardiovascular and heart disease. Their different expression in aortic tissue in patients with aortic abdominal aneurysm and their association with the progression of the disease were confirmed. They represent the potential target for the treatment of the disease. MiRNA act as biomarkers showing the potential risk of the presence of TAA, AAA and intracranial aneurysm, for the prediction of TAA and AAA progression and for the discovery of new treatment possibilities.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Patient willing and able to sign clinical trial Informed Consent
3. Patient with AAA or TAA who require an open surgical procedure, or patient with intracranial aneurysm indicated for radiological intervention

Exclusion Criteria:

1. Patient with multiorgan failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group will be made up of 50 subjects followed for the diagnosis of AAA or TAA and 20 patients with intracranial aneurysm. The control group comprises 20 subjects in total and will be made up of patients who are treated for lipid metabolism disorder
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-05-19 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The comparison of miRNA in healthy and aneurysmatic tissue | 2020 at end of trial
  miRNA will be compared in blood and in healthy and aneurysmatic tissue using ngs

CONTACTS AND LOCATIONS:
Locations (1):
- Na Homolce Hospital, Prague, Czechia